CLINICAL TRIAL: NCT02081430
Title: The Immediate Effects of Cervicothoracic Manipulation vs. Stretching on Upper Trapezius Pressure Pain Thresholds and Cervical Spine Range of Motion
Brief Title: Immediate Effects of Manipulation Versus Stretching on Upper Trapezius Pressure Pain Thresholds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNLVPT-1301
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Neurophysiological Mechanisms Manipulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CT Manipulation (Experimental): Prone cervicothoracic manipulation
  Interventions: Procedure: CT Manipulation
- Upper trapezius stretch (Active Comparator): Passive sustained stretch to upper trapezius muscle
  Interventions: Procedure: Upper trapezius stretch
- Control (No Intervention): 8 Minute wait

INTERVENTIONS:
Procedure: CT Manipulation
  Arms: CT Manipulation
Procedure: Upper trapezius stretch
  Arms: Upper trapezius stretch

SUMMARY:
The purpose of this study is to determine the immediate effects of cervicothoracic manipulation and upper trapezius stretching on upper trapezius pressure pain threshold and cervical ROM.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of current neck pain
2. Aged 18 - 70 years
3. Able to lie on stomach or back without difficulty

Exclusion Criteria:

1. 'Red flag' items indicated in Neck Medical Screening Questionnaire such as history of a tumor, bone fracture, metabolic diseases, Rheumatoid Arthritis, osteoporosis, severe atherosclerosis, prolonged history of steroid use, etc.
2. History of neck whiplash injury
3. Diagnosis from physician of cervical spinal stenosis (narrowing of spinal canal) or presence of symptoms (pain, pins and needles, numbness) down both arms
4. Presence of central nervous system involvement such as exaggerated reflexes, changes in sensation in the hands, muscle wasting in the hands, impaired sensation of the face, altered taste, and presence of abnormal reflexes
5. Evidence of neurological signs consistent with nerve root entrapment (pinched nerve in the neck)
6. Prior surgery to neck or upper back
7. A medical condition which may influence assessment of pain or pressure pain thresholds (i.e. taking analgesics, sedatives, history of substance abuse, or cognitive deficiency)
8. Diagnosis from physician of fibromyalgia syndrome
9. Currently pregnant, or could be pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Threshold | up to 10 minutes
  Using a standardized pain pressure algometer, subjects will have recordings of pressure at which onset of pain is noted

SECONDARY OUTCOMES:
Cervical Range of Motion | up to 10 minutes
  Using a CROM device, cervical spine range of motion will be measured in angular degrees

CONTACTS AND LOCATIONS:
Overall Officials: Emilio J Puentedura, PT, DPT, PhD, Principal Investigator — UNLV; William J Hanney, PT, DPT, PhD, Principal Investigator — UCF
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States